CLINICAL TRIAL: NCT03594812
Title: Effect of Aerobic Exercise Associated With Abdominal Radiofrequency on on Adipose Tissue in Women: Randomized Controlled Trial
Brief Title: Effect of Aerobic Exercise Associated With Abdominal Radiofrequency on on Adipose Tissue in Women:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Andreia Noites, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AN-007
Record Dates: First submitted 2018-07-04; First posted 2018-07-20 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2018-07

CONDITIONS: Cardiovascular Risk Factor; Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This group performed aerobic exercise just after radiofrequency therapy in the abdominal region.
  Interventions: Device: Radiofrequency; Device: Aerobic exercise
- Placebo group (Placebo Comparator): This group performed aerobic exercise just after radiofrequency therapy in the abdominal region but the radiofrequency device was switched off- Radiofrequency without power.
  Interventions: Device: Radiofrequency without power; Device: Aerobic exercise

INTERVENTIONS:
Device: Radiofrequency — Radiofrequency protocol - The radiofrequency protocol was performed in dorsal decubitus, with the head elevated at 45º. The application was in capacitive mode, with a 5 cm electrode, always in movement. The duration of the application was established in 20 minutes, maintaining the local temperature between 40ºC to 42 ºC at the epidermis.
  Arms: Experimental group
Device: Radiofrequency without power — Radiofrequency protocol - The radiofrequency protocol was performed in dorsal decubitus, with the head elevated at 45ºC (Celsius degrees). The application was in capacitive mode, with a 5 cm electrode, always in movement. The duration of the application was established in 20 minutes, maintaining the local temperature between 40ºC to 42 ºC at the epidermis. In this group, the radiofrequency device was switched off.
  Arms: Placebo group
Device: Aerobic exercise — Aerobic exercise protocol - 40 minutes of aerobic moderate-intensity exercise (45-55% of reserve heart rate) using Karvonen´s formula, performed on a cycloergometer. The duration of the exercise was divided into three parts: warm-up (from 0 to 5 minutes); body (from 5 to 35 minutes); and cooling (from 35 to 40 minutes). The entire protocol was monitored through the Polar® brand heart rate monitor and watch.

SUMMARY:
The purpose of the present study was to evaluate the effects of one session of aerobic exercise associated with radiofrequency in lipolytic activity and lipid profile.

DETAILED DESCRIPTION:
The adipose tissue is the main energetic reserve, being constituted by adipocytes, cells that accumulate lipids inside its cytoplasm, in the form of triglycerides.

Fat deposition can occur both in the subcutaneous compartment and in the visceral compartment and is the result of a positive energy balance in which there is an imbalance between the amount of calories consumed and the amount of calories expended. Thus, an excess of energy storage occurs in the form of triglycerides in adipose tissue, which results from a sedentary lifestyle and a diet based on lipid rich nutrients. When fat deposition occurs in abdominal adipose tissue may favor the development of metabolic disorders.

Recently the effectiveness of an innovative physiotherapeutic intervention - radiofrequency on adipose tissue has been studied. This therapeutic modality stimulates the lipolytic cascade, converting the triglycerides to fatty acids and glycerol. In this way, radiofrequency seems to aid in the reduction of adiposity. In addition, it assists in the reduction of the inflammatory process related to obesity, by reducing the pro-inflammatory cytokines.

The aerobic exercise, due to its low-moderate intensity, enhances the stimulation of lipolysis, by decreasing plasma insulin concentration and elevating the level of catecholamines. In this way, it influences the lipid metabolism, seeming to improve the lipid profile, through the degradation of the triglycerides as energetic substrate. In addition, the regular practice of physical exercise seems to promote a decrease in the inflammation state due to metabolic changes, through the reduction of pro-inflammatory cytokines, namely interleukin-6 and, consequently, C-reactive protein.

This study purpose understanding whether an aerobic exercise session associated with abdominal radiofrequency increases the level of lipolytic activity; To analyse the effect of four intervention sessions on abdominal adipose tissue

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Idex between 18,5 Kg/cm2 and 29,9 Kg/cm2

Exclusion Criteria:

* pregnant or intending to be in a period of an year
* participants with smoking habits
* participants with neoplasias, metabolic dysfunctions, renal pathologies, dermatological alterations
* participants with electronic devices
* participants with a condition that makes it impossible to practice physical exercise (disabling skeletal muscle pathologies and severe cardiorespiratory pathologies) participants under the effect of beta-blockers or other drugs which influence heart rate participants submitted to other fat reduce procedure

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Change in glycerol concentration | 10 minutes before the intervention and 5 minutes after the intervention
  Blood analysis collection was carried out with help from an clinical analysis technician.
Subcutaneous abdominal tissue thickness | before intervention and 2 week after (after 4 sessions of intervention )
  Measurement of the subcutaneous adipose fold by ultrasonography

SECONDARY OUTCOMES:
Change in lipid profile (LDL, HDL and triglyceride concentrations) | 10 minutes before the intervention and 5 minutes after the intervention
  Blood analysis collection was carried out with help from an clinical analysis technician.

CONTACTS AND LOCATIONS:
Locations (1):
- Andreia Noites, Porto, Portugal

REFERENCES:
- [Result] Boisnic S, Branchet MC, Birnstiel O, Beilin G. Clinical and histopathological study of the TriPollar home-use device for body treatments. Eur J Dermatol. 2010 May-Jun;20(3):367-72. doi: 10.1684/ejd.2010.0938. Epub 2010 Apr 16. PMID 20395192
- [Result] Belenky I, Margulis A, Elman M, Bar-Yosef U, Paun SD. Exploring channeling optimized radiofrequency energy: a review of radiofrequency history and applications in esthetic fields. Adv Ther. 2012 Mar;29(3):249-66. doi: 10.1007/s12325-012-0004-1. Epub 2012 Feb 29. PMID 22382873
- [Result] Goldberg DJ, Fazeli A, Berlin AL. Clinical, laboratory, and MRI analysis of cellulite treatment with a unipolar radiofrequency device. Dermatol Surg. 2008 Feb;34(2):204-9; discussion 209. doi: 10.1111/j.1524-4725.2007.34038.x. Epub 2007 Dec 17. PMID 18093200
- [Result] Hayre N, Palm M, Jenkin P. A Clinical Evaluation of a Next Generation, Non-Invasive, Selective Radiofrequency, Hands-Free, Body-Shaping Device. J Drugs Dermatol. 2016 Dec 1;15(12):1557-1561. PMID 28095578